CLINICAL TRIAL: NCT04398173
Title: A Retrospective Observational Study to Assess Prostate Cancer Detection Rate in Men Undergoing Magnetic Resonance Imaging: Comparison Between Subjects With Previous Negative Biopsy and Biopsy Naive Men
Brief Title: Detection Rate of Prostate Cancer in Men Undergoing MRI
Status: Completed | Type: Observational
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Other Study IDs: ProBiopsy-RM19
Record Dates: First submitted 2020-01-30; First posted 2020-05-21 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Prostatic Neoplasm
Keywords: magnetic resonance imaging; prostate biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (previous negative biopsy): Men with clinical suspicion of PCa, previous negative prostate biopsy who underwent prostate MRI
  Interventions: Diagnostic Test: multiparametric MRI
- Group B (biopsy naive): Men with clinical suspicion of PCa, no previous negative prostate biopsy who underwent prostate MRI
  Interventions: Diagnostic Test: multiparametric MRI

INTERVENTIONS:
Diagnostic Test: multiparametric MRI — T1-w, T2-w, diffusion weighted and dynamic contrast-enhanced imaging

SUMMARY:
To assess prostate cancer (PCa) detection rate in men undergoing magnetic resonance imaging (MRI) before planning prostate biopsy. Results will be stratified considering men with/without previous negative prostate biopsy.

Secondary objective will be to compute the negative predictive value of MRI in subject with no lesion detected at imaging or no cancer confirmed at biopsy, considering a follow-up of at least 2 years.

DETAILED DESCRIPTION:
The trial is a retrospective observational study, with the aim to compare two cohorts of patients with suspicion of PCa who will undergo MRI. Group A is composed by patients with previous negative biopsy, while group B is composed by men with no previous negative prostate biopsy.

To reach primary aim, men with positive MRI (clinically significant lesions with PI-RADS score >= 3) and biopsy data will be considered.

In men with negative MRI (clinically insignificant lesions or regions classified as PI-RADS 2 at MRI), follow-up with PSA data and repeated MRI and/or biopsy will be considered.

ELIGIBILITY:
Inclusion Criteria:

* age 50 and life expectancy greater than 10 years
* PSA values persistently greater than 4 ng/ml
* multiparametric MRI of the prostate between nov-2014 and nov-2016
* MRI with endorectal coil

Exclusion Criteria:

* previous history of PCa

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with clinical suspicion of PCa, eligible for prostate biopsy
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
PCa detection rate | 24 months
  Number of men with positive prostate biopsy over the number of men with a positive MRI

SECONDARY OUTCOMES:
Negative predictive value of MRI | 24 months
  Number of men with negative MRI or positive MRI but negative biopsy who are confirmed as negative for PCa during the follow-up over the total number of subjects considered during the follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione del Piemonte per l'Oncologia - Candiolo Cancer Institute, Candiolo, Turin, Italy